CLINICAL TRIAL: NCT05007132
Title: Prospective, Randomized, Open, Multicenter Phase II Trial to Investigate the Efficacy of Trifluridine/Tipiracil Plus Panitumumab Versus Trifluridine/Tipiracil Plus Bevacizumab as First-line Treatment of Metastatic Colorectal Cancer: FIRE-8; AIO-KRK/YMO-0519
Brief Title: Trifluridine/ Tipiracil Plus Panitumumab Versus Trifluridine/ Tipiracil Plus Bevacizumab as First-line Treatment of Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dominik Paul Modest (Other)
Responsible Party: Sponsor-Investigator, Dominik Paul Modest, Prof. Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIRE-8; 2019-004223-20 (EudraCT Number)
Record Dates: First submitted 2021-08-12; First posted 2021-08-16 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open, multicenter Phase II trial with two parallel arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Trifluridine/tipiracil, 35 mg/m² body surface area (BSA), twice daily, orally on days 1-5 and 8-12 Panitumumab at 6 mg/kg bodyweight, intravenous infusion on days 1 and 15
  Interventions: Biological: Panitumumab 20 milligram/ML; Drug: Trifluridine/Tipiracil Hydrochloride
- Arm B (Active Comparator): Trifluridine/tipiracil, 35 mg/m² body surface area, twice daily, orally on days 1-5 and 8-12 Bevacizumab at 5 mg/kg bodyweight, intravenous infusion on days 1 and 15
  Interventions: Biological: Bevacizumab; Drug: Trifluridine/Tipiracil Hydrochloride

INTERVENTIONS:
Biological: Panitumumab 20 milligram/ML — Participants receive Panitumumab at 6mg/ kg intravenously (IV) on Day 1 and 15 of each 28-day cycle. Treatment is continued until occurrence of progression according to RECIST 1.1 criteria as evaluated by the investigator or unacceptable toxicity.
  Arms: Arm A
Biological: Bevacizumab — Participants receive bevacizumab at 5 mg/ kg intravenously (IV) on Day 1 and 15 of each 28-day cycle. Treatment is continued until occurrence of progression according to RECIST 1.1 criteria as evaluated by the investigator or unacceptable toxicity.
  Arms: Arm B
Drug: Trifluridine/Tipiracil Hydrochloride — Participants receive Trifluridine/tipiracil at 35 mg/m² BSA, twice daily, orally on days 1-5 and 8-12
  Other Names: Lonsurf

SUMMARY:
FIRE-8 is a prospective, randomized, open label, multicenter phase II clinical trial. To evaluate the effecacy of trifluridine / tipiracil and panitumumab (Arm A) compared to trifluridine / tipiracil and bevacizumab (Arm B), participants will be randomly assigned to either Arm A or Arm B for the treatment of metastatic colorectal cancer.

The primary objectives of this study is to compare the effecacy of treatment with trifluridine / tipiracil plus panitumumab versus trifluridine / tipiracil plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's signed informed consent
2. Patients ≥ 18 years at the time of signing the informed consent
3. Histologically confirmed adenocarcinoma of the colon or rectum
4. Metastatic colorectal cancer (mCRC) with at least one measurable lesion according to RECIST 1.1 in a computed tomography (CT) or magnetic resonance imaging (MRI) scan performed within 5 weeks prior to randomisation
5. Metastases are primarily unresectable or patient is unable/unwilling to undergo surgery
6. RAS (Rat Sarcoma) wild-type (Kirsten rat sarcoma (KRAS), exons 2, 3, 4 and Neuroblastoma RAS viral oncogene homologue (NRAS), exons 2, 3, 4) mCRC, proven in the primary tumor or metastasis. The RAS mutational status must be determined by means of a validated test method.
7. Patient is not eligible to undergo combination chemotherapy according to investigator's assessment or unwilling to undergo combination chemotherapy.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
9. Adequate bone marrow, hepatic and renal organ function, defined by the following laboratory test results:

   * Absolute neutrophil count ≥ 1.5 x 109/L (1500/μL)
   * Hemoglobin ≥ 80 g/L (8 g/dL)
   * Platelet count ≥ 75 x109/L (75,000/μL) without transfusion
   * Total serum bilirubin of ≤ 1.5 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST/GOT) and alanine aminotransferase (ALT/GPT) ≤ 2.5 × ULN; if liver function abnormalities are due to underlying liver metastasis, AST and ALT ≤ 5 × ULN
   * Calculated glomerular filtration rate (GFR) according to Cockcroft - Gault formula or according to MDRD formula ≥ 30 mL/min or serum creatinine ≤ 1.5 x ULN
   * Urine dipstick for proteinuria < 2+ (within 14 days prior to randomisation), unless a subsequent 24-hour urine collection demonstrates < 1 g of protein in 24 hours.
10. Patients without anticoagulation need to present with an INR <1.5 x ULN and partial thromboplastin time (PTT) <1.5 x ULN. Patients with anticoagulation may be enrolled if the patient receives the medication at a stable dose for at least 2 weeks before randomisation and provided that international normalized ratio (INR) and PTT are <1.5 x ULN..
11. For females of childbearing potential (FCBP): negative pregnancy test within 14 days before randomisation and agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of <1% per year during the treatment period and for at least 6 months after the last dose of study treatment.

    A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male partner's sterilization, hormonal contraceptives that inhibit ovulation supplemented with a barrier method, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
12. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for 6 months after the last dose of study treatment. In this regard, double barrier methods are not considered to have a failure rate of < 1%. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 6 months after the last dose of study medication to avoid exposing the embryo. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Prior systemic therapy of metastatic disease. Note: Prior adjuvant chemotherapy is permitted, if completed > 3 months prior to randomisation. Multimodal treatment of rectal cancer is not considered antimetastatic therapy and does not preclude study participation
2. Known brain metastasis. In case of symptoms that are suggestive of brain metastasis, brain metastasis has to be ruled out by means of cranial CT/MRI.
3. Significant cardiovascular disease such as: New York Heart Association Class III or greater heart failure; myocardial infarction within 6 months prior to randomisation; balloon angioplasty (PTCA) with or without stenting within 6 months prior to randomisation; despite anti-arrhythmic therapy unstable cardiac arrhythmia > grade 2 NCI CTCAE; unstable angina pectoris
4. Transient ischaemic attack or cerebrovascular accident within 6 months prior to randomization, history of cerebral or aortic aneurysm or dissection
5. Medical history of deep vein thrombosis or pulmonary embolism within 6 months prior to randomisation or medical history of recurrent thromboembolic events (> 1 episode of deep vein thrombosis, pulmonary embolism, peripheral embolism) within the last 2 years.
6. Severe bleeding event within the last 6 months before randomisation (except tumor bleeding surgically treated by tumor resection)
7. Evidence of bleeding diathesis or significant coagulopathy
8. Uncontrolled hypertension defined as systolic blood pressure ≥160 mm Hg and/or diastolic ≥ 100 mm Hg under antihypertensive medication
9. Severe chronic non-healing wounds, ulcerous lesions or untreated bone fracture.
10. History of abdominal or tracheoesophageal fistula or gastrointestinal perforation, or intra-abdominal abscess -unrelated to surgery- within 6 months prior to randomisation.
11. Acute or subacute bowel obstruction, active chronic inflammatory bowel disease or chronic diarrhea
12. History of keratitis, ulcerative keratitis or severe dry eye.
13. Hypersensitivity to trifluridine/tipiracil or panitumumab or bevacizumab or any of the excipients, known hypersensitivity to Chinese hamster ovary cell products, known hypersensitivity to human or humanized antibodies
14. Current or recent (within 10 days of randomisation) use of or anticipated need for continuous treatment during study treatment with acetylsalicylic acid > 325 mg/day or treatment with dipyramidole, ticlopidine > 2 x 250 mg/day, clopidogrel > 75 mg/day, and cilostazol. Combination of these drugs are not allowed.
15. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomisation, or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 28 days prior to randomisation or anticipation of need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure
16. Core biopsy or other minor surgical procedure, excluding placement of a vascular access devices, within 3 days prior to the first dose of bevacizumab
17. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis/interstitial pneumonia, or idiopathic pneumonitis/interstitial pneumonia, or evidence of active pneumonitis or pulmonary fibrosis on screening chest imaging
18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
19. Medical history of other malignant disease than mCRC with the following exceptions:

    * patients who have been disease-free for at least three years before randomisation
    * patients with adequately treated and completely resected basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer, stage I uterine cancer
    * patients with any treated or untreated malignant disease that is associated with a 5 year survival prognosis of ≥90% and does not require active therapy
20. Known alcohol or drug abuse
21. Pregnant or breastfeeding females
22. Participation in a clinical trial or experimental drug treatment within 28 days prior to inclusion in the clinical trial or within a period of 5 half-lives of the substances administered in a clinical trial or during an experimental drug treatment prior to inclusion in the clinical trial, depending on which period is longest, or simultaneous participation in another clinical trial while taking part in this clinical trial.
23. Patient committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
24. Patient possibly dependent from the investigator including the spouse, children and close relatives of any investigator
25. Limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 36 months
  Objective response rate according to RECIST 1.1

SECONDARY OUTCOMES:
Overall survival | 36 month
  time from randomization to date of death from any cause
Progression-free survival | 36 months
  time from randomization to progression of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Sommerhauser G, Kurreck A, Stintzing S, Heinemann V, von Weikersthal LF, Dechow T, Kaiser F, Karthaus M, Schwaner I, Fuchs M, Konig A, Roderburg C, Hoyer I, Quante M, Kiani A, Fruehauf S, Muller L, Reinacher-Schick A, Ettrich TJ, Stahler A, Modest DP. Study protocol of the FIRE-8 (AIO-KRK/YMO-0519) trial: a prospective, randomized, open-label, multicenter phase II trial investigating the efficacy of trifluridine/tipiracil plus panitumumab versus trifluridine/tipiracil plus bevacizumab as first-line treatment in patients with metastatic colorectal cancer. BMC Cancer. 2022 Jul 27;22(1):820. doi: 10.1186/s12885-022-09892-8. PMID 35897060